CLINICAL TRIAL: NCT06829498
Title: HIT HEADS 2.0: Head Injury Treatment: A Randomized, Placebo-controlled, Double-blinded, Therapeutic Clinical Trial of Branched Chain Amino Acids (BCAAs) in the Treatment of Concussion
Brief Title: BCAAs in Concussion 2.0
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Akiva Cohen (Other)
Responsible Party: Sponsor-Investigator, Akiva Cohen, Researcher, Children's Hospital of Philadelphia
Organization: Children's Hospital of Philadelphia (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 23-021206
Record Dates: First submitted 2025-01-30; First posted 2025-02-17 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Concussion, Brain; Concussion, Mild; Concussion
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Drug: Branched Chain Amino Acids (Experimental): The three BCAAs will be combined together and dissolved into a flavored solution.
  Interventions: Drug: BCAA
- Placebo (Placebo Comparator): The placebo solution will have similar taste, texture, consistency and appearance as the BCAA solution.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: BCAA — The three BCAAs will be combined together and dissolved in a flavored solution.
  Arms: Drug: Branched Chain Amino Acids
Other: Placebo — The placebo solution will have similar taste, texture, consistency and appearance as the BCAA solution.
  Arms: Placebo

SUMMARY:
This study is a randomized, placebo-controlled, double-blinded, therapeutic exploratory clinical trial of branched chain amino acids (BCAAs) in the treatment of concussion. The aim of the study is to determine whether administration of high-dose BCAAs compared to placebo promotes concussion recovery.

DETAILED DESCRIPTION:
Annually, approximately 2 million concussions occur in the pediatric and young adult population. Approximately 30% of those diagnosed with concussion will experience persisting symptoms lasting beyond 28 days. Concussion is a heterogeneous injury to the brain that precipitates a complex pathophysiological process that can result in a cascade of deleterious side effects. At present, there are no targeted therapeutics that can mitigate or prevent the deleterious effects of concussion. In preclinical, analysis of ipsilateral hippocampi isolated from mice after traumatic brain injury (TBI) demonstrated that only the concentrations of the three branched chain amino acids (BCAAs) (valine, isoleucine, and leucine) were significantly reduced after injury. When these brain-injured animals received dietary supplementation with BCAAs, the concentrations of these amino acids were restored in the injured hippocampus and the injured animals demonstrated significant cognitive improvement to levels comparable to those obtained in non-injured control animals. The pilot study (NCT01860404) provides evidence of BCAAs in concussed adolescents and young adults providing a dose-response effect in reducing concussion symptoms and a return to baseline physical activity in those treated with higher total doses of BCAAs, warranting this larger trial to inform clinical practice around BCAA treatment in concussion.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females,11 - 23 years of age.
2. Weigh at least 40kg.
3. Meeting concussion criteria for the American Congress of Rehabilitative Medicine.
4. Present within 4 days of injury.
5. Post-menarchal females must have a negative urine pregnancy test and must use an acceptable method of contraception.
6. Informed consent by the participant, or for participants <18 years old both informed consent by a parent/guardian and child assent.

Exclusion Criteria:

1. Evidence of moderate or severe Traumatic Brain Injury (TBI), including Glasgow Coma Scale (GCS) <13, TBI requiring hospital admission, or TBI requiring neurosurgical intervention.
2. Prior concussion or TBI within 90 days.
3. Known history of maple syrup urine disease or known family history of maple syrup urine disease.
4. Any investigational drug use within 30 days prior to enrollment.
5. Hypersensitivity to any ingredient in the active or placebo products.
6. Participants who are pregnant, planning on becoming pregnant during the study duration, or breastfeeding.
7. Non-English speaking participants or parent/guardian.

Ages: 11 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants that have met have met criteria for recovery at 28 days post-injury, defined as return to baseline symptom levels along with feeling > 90% back to normal. | 28 days
  This will be determined by research staff at in person visits by the return to baseline symptom levels along with participant self-report of feeling > 90% back to normal. Percentage recovered at 28 days will be compared between placebo and control group by chi-square testing.

SECONDARY OUTCOMES:
Determine whether administration of high-dose BCAAs (54g/day) compared to placebo supplementation, promotes concussion recovery operationalized by the return to baseline (pre-injury) concussion symptom levels. | 28 days
  This will be determined by a comparison of total score on the Post-concussion Symptom Scale (PCSS) (22 symptoms each rated on a 0-6 Likert scale, total scale of 0-132). A participant is deemed recovered when total score is within 3 points of their pre-injury score, time to recovery will be compared among placebo and control groups by Wilcoxon rank sum test.
Determine whether administration of BCAAs leads to a lower visio-vestibular abnormality burden compared to placebo. | 28 days
  This will be determined by the visio-vestibular examination (VVE) score, a score of 0-9 based on accumulation of abnormalities on the nine elements of the VVE. Average VVE score will be compared among placebo and control groups by Wilcoxon rank sum tests.
Determine whether administration of BCAAs leads to improved pupillary light reflex (PLR) abnormalities--maximum pupil diameter compared to placebo. | 28 days
  This will be determined by a comparison of the average maximum pupil diameter (measured in mm, scale 0-9 mm) between placebo and control using Wilcoxon rank sum test, whereby larger pupil diameter represents an abnormality.
Determine whether administration of BCAAs leads to improved pupillary light reflex (PLR) abnormalities--minimum pupil diameter compared to placebo. | 28 days
  This will be determined by a comparison of the average minimum pupil diameter (measured in mm, scale 0-9 mm) between placebo and control using Wilcoxon rank sum test, whereby larger pupil diameter represents an abnormality.
Determine whether administration of BCAAs leads to improved pupillary light reflex (PLR) abnormalities-percentage of pupil constriction compared to placebo. | 28 days
  This will be determined by a comparison of the average percentage of pupil constriction change (measured in %, scale 0-100) between placebo and control using Wilcoxon rank sum test, whereby larger percent represents an abnormality.
Determine whether administration of BCAAs leads to improved pupillary light reflex (PLR) abnormalities-constriction latency compared to placebo. | 28 days
  This will be determined by a comparison of the average constriction latency (measured in ms, scale 0-1000 ms) between placebo and control using Wilcoxon rank sum test, whereby shorter latency represents an abnormality.
Determine whether administration of BCAAs leads to improved pupillary light reflex (PLR) abnormalities-average constriction velocity compared to placebo. | 28 days
  This will be determined by a comparison of the median average constriction velocity (measured in mm/s, scale 0-5 mm/s) between placebo and control using Wilcoxon rank sum test, whereby faster constriction velocity represents an abnormality.
Determine whether administration of BCAAs leads to improved pupillary light reflex (PLR) abnormalities--peak constriction velocity compared to placebo. | 28 days
  This will be determined by a comparison of the average peak constriction velocity (measured in mm/s, scale 0-5 mm/s) between placebo and control using Wilcoxon rank sum test, whereby faster constriction velocity represents an abnormality.
Determine whether administration of BCAAs leads to improved pupillary light reflex (PLR) abnormalities-average dilation velocity compared to placebo. | 28 days
  This will be determined by a comparison of the median average dilation velocity (measured in mm/s, scale 0-5 mm/s) between placebo and control using Wilcoxon rank sum test, whereby faster dilation velocity represents an abnormality.
Determine whether administration of BCAAs leads to improved pupillary light reflex (PLR) abnormalities-peak dilation velocity compared to placebo. | 28 days
  This will be determined by a comparison of the average peak dilation velocity (measured in mm/s, scale 0-5 mm/s) between placebo and control using Wilcoxon rank sum test, whereby faster velocity represents an abnormality.
Determine whether administration of BCAAs leads to improved pupillary light reflex (PLR) abnormalities-T75 compared to placebo. | 28 days
  This will be determined by a comparison of the average time to reach 75% of the original baseline pupil diameter (T75) after peak constriction (measured in s, scale 0-4 s) between placebo and control using Wilcoxon rank sum test, whereby faster time represents an abnormality.
Determine whether administration of BCAAs leads to subjective improvement in sleep quality compared to placebo. | 28 days
  Sleep quality will be determined by utilization of the PROMIS sleep questionnaire with 8 questions and a 5 point scale (1- not at all, 2- a little bit, 3- somewhat, 4- quite a bit and 5- very much). The PROMIS Sleep Disturbance score is calculated by adding up the raw scores for each item on the PROMIS Sleep Disturbance scale. The score is then rescaled to a standardized T-score using a conversion table. A higher score indicates greater sleep disturbance. Total range of score is 8-40. Average score will be compared between placebo and control using Wilcoxon rank sum test.
Determine whether administration of BCAAs leads to subjective improvement in physical activity compared to placebo. | 28 days
  Physical activity will be determined by utilization of the PROMIS sleep questionnaire with 8 questions and an aggregate score of X. Physical activity will be determined by utilization of the PROMIS Physical Activity questionnaire with 8 questions and a 5 point scale (1- not at all, 2- a little bit, 3- somewhat, 4- quite a bit and 5- very much). A higher aggregate score may be indicative of greater activity limitations or reduced activity levels. Total range of score is 8-40. Average score will be compared between placebo and control using Wilcoxon rank sum test.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Corwin, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Corwin DJ, Myers SR, Arbogast KB, Lim MM, Elliott JE, Metzger KB, LeRoux P, Elkind J, Metheny H, Berg J, Pettijohn K, Master CL, Kirschen MP, Cohen AS. Head Injury Treatment With Healthy and Advanced Dietary Supplements: A Pilot Randomized Controlled Trial of the Tolerability, Safety, and Efficacy of Branched Chain Amino Acids in the Treatment of Concussion in Adolescents and Young Adults. J Neurotrauma. 2024 Jun;41(11-12):1299-1309. doi: 10.1089/neu.2023.0433. Epub 2024 Apr 11. PMID 38468511